CLINICAL TRIAL: NCT06461442
Title: Efficacy and Safety of Cryotherapy Versus 5-Fluorouracil in the Treatment of Actinic Keratosis: A Prospective, Randomized Controlled, Intra-Individual Trial
Brief Title: Efficacy and Safety of Cryotherapy Versus 5-Fluorouracil in the Treatment of Actinic Keratosis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2164169
Record Dates: First submitted 2024-06-10; First posted 2024-06-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Actinic Keratoses
Keywords: cryotherapy; 5-Fluorouracil
MeSH Terms: conditions — Keratosis, Actinic | interventions — Cryotherapy; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cryotherapy and 5-Fluoruracil (Experimental): Each actinic keratosis lesion, or treatment area, will be randomly assigned to receive either cryotherapy or 5-fluoruracil treatment.
  Interventions: Procedure: Cryotherapy; Drug: 5Fluorouracil

INTERVENTIONS:
Procedure: Cryotherapy — Extremely cold liquid (liquid nitrogen) will used by a dermatologist to freeze and destroy abnormal cells in the treatment areas randomized to this treatment.
Drug: 5Fluorouracil — Patients will apply 5% 5-Fluorouracil cream in a thin layer twice daily for 4 weeks on the treatment areas randomized to this treatment.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness and safety of two treatments-cryotherapy and 5-Fluorouracil (5-FU)-for actinic keratosis, a common skin condition caused by long-term sun exposure. Cryotherapy is a treatment that uses extreme cold produced by liquid nitrogen to freeze and destroy abnormal cells, and 5-FU is a topical cream applied to the skin to treat lesions by interfering with cell growth. The main questions this trial aims to answer are:

* Which treatment, cryotherapy or 5-FU, is more effective in reducing the number of actinic keratosis lesions?
* What are the side effects associated with each treatment?
* How do these treatments impact patient satisfaction, cosmetic outcomes, and health-related quality of life?

Participants will:

* Undergo a baseline assessment where their demographics information such as age, sex, race, smoking status, and medical history are recorded, along with the number and severity of actinic keratosis lesions.
* Receive both cryotherapy and 5-FU, with each treatment applied to different areas of their body. The area of the body to receive each treatment is decided by a random process (like flipping a coin).
* Complete weekly surveys to monitor for side effects during and after the treatment period.
* Return to the clinic for follow-up assessments at 3 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has a clinical diagnosis of 10 or more AKs in the head, neck, or extremities areas
* Able to give informed consent themselves
* Willing to return for follow up visits

Exclusion Criteria:

* Cognitively Impaired
* Incarcerated
* Non-English speakers
* Immuno-comprised status
* Received any kind of treatment for AK within the past 2 months
* Use of systemic retinoids within the past 3 months
* Suspicion of cancer in the target area
* Porphyria
* Genetic skin cancer disorders
* Allergy to trial drugs or peanut/soy products
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Partial clearance rate | 3 months and 12 months
  Proportion of patients with at least a 75% reduction in the number of baseline AK lesions within the selected treatment area

SECONDARY OUTCOMES:
Complete clearance rate | 3 months and 12 months
  Proportion of patients with no clinically visible AK lesions (i.e., a 100% reduction in the number of baseline AK lesions) within the selected treatment area
Percent reduction of AK lesions | 3 months and 12 months
  Decrease in number AK lesions from baseline within the selected treatment area
Rate of progression to keratinocyte carcinoma | 3 months and 12 months
  Proportion of AK lesions within the treatment area that progress to keratinocyte carcinoma
Recurrence rate | 3 months and 12 months
  Proportion of participants with recurrent or new lesions within the treatment area
Patient satisfaction | 3 months and 12 months
  Proportion of patients who would choose the same treatment again and if they would recommend it to others
Health-Related Quality of Life | 3 months and 12 months
  Skindex-29 questionnaire
Cosmetic outcome | 3 months and 12 months
  The cosmetic outcome will be evaluated using a 4-point scale (1 = excellent, 2 = good, 3 = moderate, and 4 = poor) by an investigator who is blinded to the treatment allocation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — UC Davis Department of Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

REFERENCES:
- [Background] Jansen MHE, Kessels JPHM, Nelemans PJ, Kouloubis N, Arits AHMM, van Pelt HPA, Quaedvlieg PJF, Essers BAB, Steijlen PM, Kelleners-Smeets NWJ, Mosterd K. Randomized Trial of Four Treatment Approaches for Actinic Keratosis. N Engl J Med. 2019 Mar 7;380(10):935-946. doi: 10.1056/NEJMoa1811850. PMID 30855743